CLINICAL TRIAL: NCT01213186
Title: Phase 2 Study of UC-MSC in Restoring CD4 T Cell Counts and Reducing Immune Activation in HIV-infected Patients Underlying Long-term Antiviral Therapy: a Multicenter, Does-escalating, Randomized, Double-blind, Controlled Trial.
Brief Title: Umbilical Cord Mesenchymal Stem Cells for Immune Reconstitution in HIV-infected Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu-Sheng Wang (Other)
Responsible Party: Sponsor-Investigator, Fu-Sheng Wang, Director, Beijing 302 Hospital
Organization: Beijing 302 Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: beijing302-001
Record Dates: First submitted 2010-09-28; First posted 2010-10-01 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Human Immunodeficiency Virus; Disorder of Immune Reconstitution
Keywords: stem cell; hiv; CD4; immune activation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drug: high dose of MSC treatment (Experimental): Participants will receive high dose of MSC from Day 0 through the Week 48 study visit. Participants will then be followed until the Week 48 study visit.
  Interventions: Drug: high dose of MSC
- low dose of MSC treatment (Experimental): Participants will receive a low dose of MSC treatment from Day 0 through the Week 48 study visit, and then follow-ed up for additional 48 weeks.
  Interventions: Drug: low dose of MSC treatment
- low dose of MSC (Placebo Comparator): Participants will receive a saline placebo treatment from Day 0 through the Week 48 study visit, and then follow-ed up for additional 48 weeks.

INTERVENTIONS:
Drug: high dose of MSC — Taken i.v., at week 0, 4, 12, 24, 36 and 48, at a dose of 1.5*10E6/kg for 48 weeks.
  Other Names: MSC treatment dose
  Arms: Drug: high dose of MSC treatment
Drug: low dose of MSC treatment — Taken i.v., at week 0, 4, 12, 24, 36 and 48, at a dose of 0.5*10E6/kg for 48 weeks.
  Other Names: MSC low dose
  Arms: low dose of MSC treatment

SUMMARY:
HIV-1 infection is characterized by progressive depletion of CD4+ T cells that eventually leads to clinically significant immunodeficiency. A chronic generalized immune activation is now being recognized to be the main driving force for T cell depletion, loss of anti-HIV-1 immunity and disease progression during chronic HIV-1 infection. However, it is still unknown whether reducing immune activation will restore CD4 T cell counts and leading to immune reconstitution in chronic HIV infection. Mesenchymal stem cells (MSC) have been demonstrated to decrease immune responses of the host, and can suppress inflammation in HIV-infected non-responders. Here, the investigators propose a hypothesis that MSC can reduce immune activation which subsequently lead to the restoration of CD4 T-cell counts dependent on dose of transfused MSCs in HIV-infected patients.

DETAILED DESCRIPTION:
Although HIV-1 infection is characterized by progressive depletion of CD4+ T cells that eventually leads to clinically significant immunodeficiency, a chronic generalized immune activation is now being recognized to be the main driving force for T cell depletion, loss of anti-HIV-1 immunity and disease progression during chronic HIV-1 infection. In particular, this immune activation has been identified as a disease determinant independent of viral load or cell death in HIV-1 infection. A series of clinical evidences have indicated that activated CD8 T cells may attack body cells infected with viruses. Because of this, CD4 cells infected with HIV are frequently destroyed by CD8 cells.

Mesenchymal stem cells (MSCs) are the adult stem cells originating from the mesenchymal and connective tissue of bone marrow, adipose tissue, placenta, umbilical cord, cord blood, peripheral blood, liver, etc. These cells show immunomodulation, self-renewal, and multi-directional differentiation potential. In particular, MSCs have recently emerged as promising candidates for cell-based immunotherapy because they can modulate the immune response in various ways. A series of studies have indicated that secretion of dissoluble cytokines and direct contact with MSCs can block the development and functioning of antigen-presenting cells, inhibit the differentiation of B cells, and suppress the immune response of T cells and natural killer cells. The immunosuppressive effect of infused MSCs has been successfully employed in the treatment of acute severe graft-versus-host disease (GVHD). Thus, MSC may reduce inflammatory responses and promote tissue recovery in human diseases.

The purpose of this study is to learn what dose of transfused MSC reduces the level of activation of CD8 cells in people infected with HIV. The decreased activation of CD8 cells may lead to a more CD4 T cell restoration in HIV infection. This study will also look at what dose of MSCs is tolerated and its safety in HIV- infected patients.

Participants in this study will be randomly assigned to one of three treatment arms:

Arm A:Participants will receive 48 weeks of low dose of MSC treatment followed by 48-week follow-up observation.

Arm B:Participants will receive 48 weeks of high dose of MSC treatment followed by 48-week follow-up observation.

Arm C: Participants will receive 48 weeks of saline placebo followed by 48-week follow-up observation.

Study treatment will be given at 0, 4, 12, 24, 36 and 48 week since the onset of treatment. There will be an additional 48 weeks of follow-up for purposes of safety. After treatment has started, participants will be asked to come to the clinic on Weeks 4, 12, 24, 36, 48,60,72,84 and 96. At each visit participants will receive enough study treatment to last until the next visit. Each visit will last between 2 and 3 hours. At most visits participants will have a physical exam, answer questions about any medications they are taking and how they are feeling, and have blood drawn for safety to assess CD4/CD8 cell counts and viral load. Some additional blood will also be stored for immunology testing. At some visits participants will be asked questions about their medication and medical history, have pupils dilated, have a hearing test, and have an electrocardiogram (EKG). Some visits will require participants to arrive fasting. Pregnancy tests may also be conducted if the participant is able to become pregnant or if pregnancy is suspected.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infected
2. antiretroviral therapy (ART) for at least 24 months prior to study entry and continue within the 24 months after study entry
3. CD4 count less than or equal to 250 cells/mm3 continuously and more than 50 cells/mm3 before entry and at screening, obtained within 30 days prior to study entry
4. Viral load less than or equal to 50 copies/mL obtained within 30 days prior to study entry
5. Certain specified laboratory values obtained within 30 days prior to study entry. More information on this criterion can be found in the study protocol.
6. Documentation that pre-entry specimen for the primary immune activation endpoint responses has been obtained
7. No history of CDC category C AIDS-related opportunistic infections
8. Karnofsky performance score greater than or equal to 70 within 30 days prior to study entry
9. Ability and willingness to provide informed consent

Exclusion Criteria:

1. coinfection with other virus, including serum HCV RNA positive, or one of followings are positive in antiHAV/anti-HDV/anti-HEV plus ALT more than 80 IU/L.
2. history of combination with other severe diseases including renal, circulatory, respiratory, digestive, endocrine, neural and immunological diseases and tumors.
3. WBC <2.5*10E9/L, platlet counts <50*10E9/L, Hb <80g/L, lactate >2 mmol/L;
4. allergic constitution;
5. Accepting other immunomodulatory drugs within 6 months prior screening.
6. drug addiction;
7. other conditions possibly influencing the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
the total CD4 T cell counts compared with CD4 T cell counts at baseline | At Baseline and at week 4, 12, 24, 36,48,60,72,84,96

SECONDARY OUTCOMES:
the CD38 expression on CD8 T cells | At Baseline and at week 4, 12, 24, 36,48,60,72,84,96
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at baseline and up to week 96
plasma RNA copies/mL | At Entry and at Weeks 24, 48, 72, 96
the ratio of CD4 and CD8 T cells | At Baseline and at week 4, 12, 24, 36,48,60,72,84,96
the HLA-DR expression on CD8 T cells | At Baseline and at week 4, 12, 24, 36,48,60,72,84,96
Quality of live | At Baseline and at week 4, 12, 24, 36,48,60,72,84,96
the occurring rate of tumor | At Baseline and at week 24, 48, 72, 96
occurring rate of opportunistic infections | At Baseline and at week 24, 48, 72, 96

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Professor, Principal Investigator — Beijing 302 Hospital
Locations (3):
- China (3):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - Xinjiang Hospital of Infectious Diseases, Ürümqi, Xinjiang
  - the Yunnan Hospital of Infectious Diseases, Kunming, Yunnan

REFERENCES:
- [Background] Appay V, Sauce D. Immune activation and inflammation in HIV-1 infection: causes and consequences. J Pathol. 2008 Jan;214(2):231-41. doi: 10.1002/path.2276. PMID 18161758
- [Background] Uccelli A, Moretta L, Pistoia V. Mesenchymal stem cells in health and disease. Nat Rev Immunol. 2008 Sep;8(9):726-36. doi: 10.1038/nri2395. PMID 19172693
- [Derived] Zhang Z, Fu J, Xu X, Wang S, Xu R, Zhao M, Nie W, Wang X, Zhang J, Li T, Su L, Wang FS. Safety and immunological responses to human mesenchymal stem cell therapy in difficult-to-treat HIV-1-infected patients. AIDS. 2013 May 15;27(8):1283-93. doi: 10.1097/QAD.0b013e32835fab77. PMID 23925377